CLINICAL TRIAL: NCT04721054
Title: Thoracic Epidural Versus General Anesthesia for Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Thoracic Epidural Versus General Anesthesia for Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, arshad khushdil, Assistant Professor, Armed Forces Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 104589
Record Dates: First submitted 2021-01-02; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Epidural Anesthesia; General Anesthesia
Keywords: headache; blood pressure
MeSH Terms: conditions — Headache | interventions — Cholecystectomy, Laparoscopic; Bupivacaine; Lidocaine

STUDY DESIGN:
Intervention Model Description: one group to be studied for effects of epidural anesthesia and other group for effects of general anesthesia
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group receiving thoracic epidural anesthesia (Active Comparator)
  Interventions: Drug: Thoracic epidural effect on heart rate in Laparoscopic Cholecystectomy (bupivacaine and lignocaine)
- group receiving thoracic general anesthesia (Active Comparator)
  Interventions: Drug: general anesthesia effect on heart rate in Laparoscopic Cholecystectomy

INTERVENTIONS:
Drug: Thoracic epidural effect on heart rate in Laparoscopic Cholecystectomy (bupivacaine and lignocaine) — patients in epidural anesthesia were given epidural anesthesia and assessed for heart rate and mean arterial pressure
  Other Names: Thoracic epidural effect on mean arterial pressure in Laparoscopic Cholecystectomy
  Arms: group receiving thoracic epidural anesthesia
Drug: general anesthesia effect on heart rate in Laparoscopic Cholecystectomy — patients in general anesthesia were given epidural anesthesia and assessed for heart rate and mean arterial pressure
  Other Names: general anesthesia effect on mean arterial pressure in Laparoscopic Cholecystectomy
  Arms: group receiving thoracic general anesthesia

SUMMARY:
Eighty two patients planned to undergo elective laparoscopic cholecystectomy were divided into two groups, T and G, randomly. In Group T all patients underwent laparoscopic cholecystectomy under thoracic epidural anesthesia with 12mlof 0.25% bupivacaine and 1% lignocaine plain whereas in group G all patients underwent surgery under general anesthesia. Intra-operative heart rate, mean arterial pressure (MAP) and post operative opioid consumption in first 24hrs were recorded as primary outcomes whereas presence or absence of respiratory complication and duration of hospital stay as secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. patients having ASA statusI-III
2. age more than 18 years,
3. both genders
4. planned to undergo laparoscopic cholecystectomy

Exclusion Criteria:

1. Patients who did not give consent,
2. Allergic to local anesthetic
3. Hemodynamically unstable,
4. Pregnant, full stomach patients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
effectiveness of thoracic epidural anesthesia with general anesthesia for Laparoscopic cholecystectomy in terms of change in heart rate during surgery in immediate 24 hours-heart rate. | changes in heart rate at 24 hours of surgery.
  the efficacy of thoracic epidural anesthesia was compared with general anesthesia for laproscopic cholecystectomy in the immediate post operative period in terms of intra operative heart rate.
effectiveness of thoracic epidural anesthesia with general anesthesia for Laparoscopic cholecystectomy in terms of change in mean arterial blood pressure during surgery in immediate 24 hours-mean arterial blood pressure. | changes in mean arterial pressure at 24 hours of surgery
  efficacy of thoracic epidural anesthesia was compared with general anesthesia for laproscopic cholecystectomy in the immediate post operative period in terms of mean arterial blood pressure intra operatively and in immediate post operative period

CONTACTS AND LOCATIONS:
Locations (1):
- Military Hospital, Rawalpindi, Punjab Province, Pakistan